CLINICAL TRIAL: NCT04925245
Title: Clinical Reminder to Improve Appropriateness of Echocardiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Paul A. Heidenreich, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CSRPecho1
Record Dates: First submitted 2019-08-19; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Echocardiography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Reminder (Experimental)
  Interventions: Other: Clinical Reminder
- No Reminder (No Intervention)

INTERVENTIONS:
Other: Clinical Reminder — Clinical reminder in the electronic medical record
  Arms: Clinical Reminder

SUMMARY:
This study will test a clinical reminder to show recent echocardiograms when a new echocardiogram is ordered. The goal is to avoid unnecessary comprehensive echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Echo ordered

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1365 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Comprehensive echo ordered | 24 hours from when when the initial order was placed
  Number of comprehensive echos completed

SECONDARY OUTCOMES:
Cost of Echocardiography | 30 days
  Cost of echocardiography during the hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No